CLINICAL TRIAL: NCT02117180
Title: Evaluation of the Nutritional Adequacy of a Diet Low in Fermentable Oligosaccharides, Disaccharides, Monosaccharides and Polyols (FODMAP's) in Children With Functional Gastrointestinal Disorders.
Brief Title: Nutritional Adequacy of a FODMAP Diet in Children
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Anne Payne (Other)
Collaborators: University of London (Other)
Responsible Party: Sponsor-Investigator, Dr Anne Payne, Associate Professor/Academic Lead for Nutrition & Dietetics, University of Plymouth
Organization: University of Plymouth (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CdeK2014
Record Dates: First submitted 2014-04-09; First posted 2014-04-17 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Functional Gastrointestinal Disorders in Children
Keywords: functional gastrointestinal disorders; FGID; children; FODMAP
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FODMAP's diet (Other): A diet low in Fermentable Oligosaccharides, Disaccharides, Monosaccharides And Polyols (FODMAPs)
  Interventions: Other: FODMAP's diet

INTERVENTIONS:
Other: FODMAP's diet — The safety and efficacy of a low FODMAP diet will be evaluated in a convenience sample of children with functional gastrointestinal disorders, over a 6 week intervention period.

SUMMARY:
This pilot study aims to establish whether a low FODMAP diet is safe in children with functional gastrointestinal disorders. The practicality of implementing this diet will be evaluated as well as symptom improvement and quality of life. A larger intervention trial, if deemed appropriate, will then follow to assess symptom efficacy in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 10-16 years
* Informed consent and assent obtained
* Patients with diagnosed FGID according to Rome III criteria: i.e. category H2b (irritable bowel syndrome) and H2d (childhood functional abdominal pain)

Exclusion Criteria:

* Patients with other gastrointestinal conditions (e.g. coeliac disease, inflammatory bowel disease)
* Patients with food allergies
* Patients with a weight for age below -2 Standard Deviations (SD) (below 0.4th centile) on the UK WHO growth charts.
* Patients with known micronutrient deficiencies determined by blood levels prior to study
* Patients without informed consent and assent obtained

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Energy and nutrient intake | Baseline, 6 weeks
  Energy and nutrient intake will be assessed using a 4-day estimated food diary at baseline and 6-weeks after dietary intervention. Comparison will be made between baseline and 6-week data and with United Kingdom (UK) Reference Nutrient Intakes.

SECONDARY OUTCOMES:
Practicality of the FODMAP diet; impact of diet on Functional Gastro-Intestinal .Disorders (FGID) symptoms and stools | Baseline, 6 weeks
  Practicality of the FODMAP diet will be evaluated using a standardised structured questionnaire.
  The impact of a low FODMAP diet on FGID symptoms and stools will be assessed using a validated symptom questionnaire and the Bristol Stool Chart.
  The impact of a low FODMAP diet on quality of life will be assessed using the Pediatric Quality of Life Inventory (PedsQL) Gastrointestinal Symptoms Module.
Anthropometry: weight and mid-arm circumference | Baseline, 6 weeks
  Anthropometric measurements will be taken at baseline and 6 weeks after dietary intervention. Comparison will be made between baseline and 6-week data for weight and mid upper arm circumference, as well as comparing both baseline and 6-week data to the UK-WHO growth standards.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Payne, PhD, Study Director — University of Plymouth; Claire de Koker, BSc (Hons), Principal Investigator — Chelsea and Westminster NHS Foundation Trust, UK
Locations (1):
- Chelsea and Westminster NHS Foundation Trust, London, United Kingdom